CLINICAL TRIAL: NCT06003855
Title: Oxygen-guided Supervised Exercise Therapy in Peripheral Artery Disease
Brief Title: Oxygen-guided Supervised Exercise Therapy
Acronym: MOMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E4632-P
Record Dates: First submitted 2023-07-25; First posted 2023-08-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral arterial disease; atherosclerosis; arterial occlusive disease; gait
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: Two groups will complete 12 weeks (36 sessions) of supervised exercise therapy. One group will complete the standard of care and the other group will complete the muscle oxygen guided supervised exercise therapy. Subjects will be randomly assigned to one of the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen guided supervised exercise (Experimental): Modified-SET parameters will be determined from resting StO2 during 10 minutes of sitting. The StO2 threshold will be set at 15% lower than baseline StO2 levels. After warm-up, the subjects will walk until they reach the StO2 threshold. The subjects will be instructed to stop walking once they reach the threshold and to rest until the StO2 level returns to the baseline level. Then, subjects will be instructed to begin walking again and this cycle will be repeated for 50 total minutes. The threshold was selected to be above the 31% drop associated with claudication onset time. If subjects experience pain earlier than the 15% drop, the threshold will be progressively decreased by 5%, as needed. Subjects will repeat this for up to 50 minutes (including walking and rest). Walking speed and treadmill incline will be adjusted to allow for 5-10 minutes of walking before reaching the threshold. Subjects will complete 3 sessions/week for 12 weeks.
  Interventions: Behavioral: Supervised exercise therapy
- Standard supervised exercise (Active Comparator): After the warmup, subjects will walk until claudication pain becomes severe and needs to stop. Then subjects will rest until claudication pain subsides. Afterwards, subjects will walk again, repeating the cycle for up to 50 minutes (including walking and rest). Walking speed and treadmill incline will be adjusted during the SET session to allow individuals with PAD to walk for 5-10 minutes before claudication symptoms arise. Time at each speed and incline, along with rest times will be recorded during each exercise session. Subjects will complete 3 sessions/week for 12 weeks.
  Interventions: Behavioral: Supervised exercise therapy

INTERVENTIONS:
Behavioral: Supervised exercise therapy — Subjects will be enrolled in a 12-week intervention program of either modified supervised exercise therapy or standard supervised exercise therapy. The program will be 3 sessions/week for 12 weeks. Each session will consist of 50 minutes plus 5 minutes warm up and cool down.

SUMMARY:
Peripheral artery disease (PAD) is a cardiovascular disease manifesting from systemic atherosclerosis, which blocks the leg arteries and results in insufficient blood flow to the lower extremities. Limb ischemia from PAD is the most common disorder treated within the vascular surgery service at the Omaha Veterans' Affairs Medical Center. PAD also accounts for one-third of the operations performed in the VA Medical Centers nationwide. This project aims to establish the feasibility and acceptability of a muscle oxygen-guided supervised exercise program for patients with PAD. The investigators will determine the potential benefits of using this intervention over standard supervised exercise therapy. This modified intervention may enable patients to increase overall physical activity without the negative impacts on muscle structure and function. Increasing physical activity will decrease cardiovascular morbidity and mortality. If proven beneficial, the findings will lead to an improved exercise program that directly benefits veterans nationwide.

DETAILED DESCRIPTION:
The long-term goal of this research is to improve mobility, functional independence, and quality of life in patients with peripheral artery disease (PAD) by developing conservative interventions. PAD is a manifestation of atherosclerosis, which produces blockages in the leg arteries, and results in insufficient blood flow to the legs. PAD results in significant gait deficits and an overall sedentary lifestyle. The investigators' prior work showed that the biochemical (oxidative stress and mitochondrial dysfunction) and histological (myofiber degeneration and fibrosis) characteristics of PAD muscles are altered compared to controls. These myopathic changes are due to cycles of ischemia and reperfusion, and they correlate to functional limitations (walking distance and calf muscle strength). Limb ischemia from PAD is the most common disorder treated within the vascular surgery service of the Omaha Veterans Affairs Medical Center. The most effective treatment for increasing the distances that patients with PAD can walk is supervised exercise therapy (SET). However, SET uses pain onset to guide exercise intensity and rest cycles. These repeated bouts of ischemia/reperfusion could cause further pathological damage to muscle myofibers and oxidative processes. Such adverse effects of ischemia may explain why not all patients improve with SET. Preventing cycles of ischemia-reperfusion during SET can improve walking performance without further muscle biochemistry damage in patients with PAD. The investigators propose using hemodynamic responses to modulate exercise intensity and prevent ischemia during SET. Muscle oxygen-guided supervised exercise therapy (M-SET) can prevent ischemia onset and thus preserve muscle mass and function during exercise therapy in patients with PAD. The aims are:

Aim 1: To determine the exercise outcomes of an M-SET versus a standard SET session in patients with PAD. Aim 2: To determine the acute effect of M-SET versus standard SET on oxidative stress and inflammation in patients with PAD. Aim 3: To determine the effect of 12 weeks of M-SET versus standard SET on exercise outcomes, muscle biochemistry, and subject-reported preference in patients with PAD.

The investigators will measure exercise outcomes during one session each of M-SET (using StO2 on the calf to modulate exercise) and SET, in 12 patients with PAD using a cross-over design. Exercise outcomes will be assessed by the total distance patients walked during the session, metabolic cost, metabolic equivalents of the task, physical activity enjoyment, and rate of perceived exertion. In Aim 2, oxidative stress will be measured using peripheral blood mononuclear cells before and after each exercise session (SET and M-SET) in all patients. During the standard SET session, subjects will walk until claudication pain becomes severe and the participant needs to stop. Then subjects will rest until claudication pain subsides. Afterward, subjects will walk again, repeating the cycle for up to 50 minutes. M-SET will use an StO2 threshold that is 15% lower level than baseline StO2 levels. Subjects will stop walking once they reach the threshold and rest until StO2 levels return to baseline. Then, subjects will begin walking again, repeating this cycle for 50 total minutes (including walking and rest). Patients from Aims 1 and 2 will be randomly assigned to either a 12-week M-SET or standard SET (6 per group) program. Training will be performed three times weekly as described above. Subjects will be evaluated before and after the intervention to capture initial and absolute walking distances and 7-day physical activity. Muscle biochemistry will be quantified using mitochondrial function, mitochondrial oxidative dynamics, and reactive oxygen species production before and after training. Results will support a full clinical trial and rehabilitation recommendations.

ELIGIBILITY:
Inclusion Criteria:

At entry into the study, all subjects must:

* Be able to give written, informed consent
* Have documented lower extremity arterial occlusive disease based on ankle/brachial index measurements and/or arterial imaging
* Demonstrate positive history of chronic claudication
* Have a stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks

Exclusion Criteria:

Any potential subjects will be excluded if they have:

* Rest pain or tissue loss due to PAD (Fontaine stage III and IV)
* Acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma
* Walking capacity limited by conditions other than claudication including leg (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Distance walked | Before and after 12 week exercise program
  Total distance walked during the exercise session (standard or M-SET) will be determined using the total time of walking multiplied by the walking speed.
Energy expenditure | Before and after 12 weeks after the exercise program
  Energy expenditure57 will be assessed via oxygen consumption as measured by a metabolic cart (K5, Cosmed USA, Inc., Chicago, IL). Subjects will stand quietly for five minutes to collect resting energy expenditure. Standing steady state energy expenditure will be calculated for each subject by plotting VO2 and assigning a sliding best fit line over a two-minute window. Steady-state oxygen consumption in ml/kg/min will be calculated during the exercise session. Energy cost of transport will be calculated by subtracting the energy consumption values at standing from walking to achieve net metabolic cost for each bout of exercise.
Reactive oxygen species | Before exercise, immediately after exercise, 30 minutes after exercise, and 1 hour after exercise
  Quantification of reactive oxygen species (ROS) related markers and free radicals: Electron paramagnetic resonance (EPR), which has been known as a gold standard for free radical assessment, will be used to quantify free radicals such as superoxide as we have previously performed (1-3). Plasma samples will be used for measuring ROS-related markers such as TAC, SOD, GSH:GSSG, ONOO- and MDA with commercially available and previously validated ELISA Assay Kits (CAT#s ab65329, ab65354, ab138881, ab233469, and ab233471 Abcam, UK) according to the manufacturer's instructions60. The average intra-assay variability measured as the coefficient of variation for each sample was 2.9%, 3.8%, and 3.3% for SOD, TAC, and MDA, respectively.
Protein expression of ROS-related enzymes | Before exercise, immediately after exercise, 30 minutes after exercise, and 1 hour after exercise
  Protein expression of ROS-related enzymes: Enzymes related to ROS will be quantified with western blots of isolated PBMCs analyzed for catalase, 4 hydroxynonenal (4HNE), and glutathione peroxidase 1 (GPX) (4). All samples will be homogenized in RIPA buffer (Boston Bioproducts) and 100X protease inhibitor (Sigma Aldrich). A 150-volt electrical potential will be applied to the gel for 1 hr to separate proteins based on mass. A 250-volt electrical potential will then be applied to the gel for 7 min to transfer protein bands to transfer paper with TurboTransfer (Biorad). Primary antibodies for catalase, 4HNE, and GPX will be recombinant anti-catalase antibody (ab209211), anti-4 hyroxynonenal antibody (ab243070), and recombinant anti-glutathione peroxidase 1 antibody (ab108429), respectively.
Markers of systemic inflammation | Before exercise, immediately after exercise, 30 minutes after exercise, and 1 hour after exercise
  Markers of systemic inflammation: Standard ELISA kits will be used to test blood samples for interleukin 6, tumor necrosis factor-a, vascular cell adhesion protein 1, and vascular endothelial growth factor-a (Cat#s, ab178013, ab285312, ab223591, ab119566). Oxidized low density lipoproteins (LDL) will be measured with an oxidized LDL assay kit (ab242302). All measurements will be made per validated manufacturer specifications.
Initial and absolute walking distances | Before and after 12 week supervised exercise program
  Initial and absolute walking distances will be determined from the progressive-load treadmill test. Subjects will walk on a treadmill that starts at 0% grade and 2.0 mph. Every two minutes, the grade will be increased by 2% up to a maximum of 15% grade, and the speed held constant throughout the test. Initial claudication distance is the distance walked prior to claudication pain onset. Absolute claudication distance is the total distance walked before subjects had to stop walking due to claudication pain.
Comprehensive mitochondrial respiratory complex function | Before and after 12 week supervised exercise program
  Comprehensive mitochondrial respiratory complex function (complex I, II, III, IV, and V) will be completed with previously validated high resolution respirometry with complex agonists/antagonists. Skeletal muscle tissue will be manually teased and permeabilized with 15 l of digitonin for 30 min. Samples will then be rinsed twice in 2 ml of MIRO5 for 10-min. 3-5 mg (dry weight) of tissue will then be isolated and placed in the high-resolution respirometer with 2 ml of MIRO5 solution. The order and quantity of each agonist and antagonist will be applied as follows: 5 l malate and 10 l glutamate (complex I agonist), 20 l adenosine diphosphate (complex V agonist), 20 l succinate (complex II agonist), 1 l rotenone (complex I antagonist), 1 l oligomycin (complex V antagonist), 1 l antimycin A (complex III antagonist), and 5 l ascorbate + 5 l TMPD (complex IV agonist).
Mitochondrial dynamics | Before and after 12 week supervised exercise program
  Specific proteins we will assess are Fis-1 and DRP-1 (fission), Mfn-1, Mfn-2 and OPA-1 (fusion), and UPC-1 and UCP-2 (dynamics). We will perform the same Western Blot technique mentioned in Aim #262. Primary antibodies for Fis-1, DRP-1, Mfn-1, Mfn-2, OPA-1, UPC-1, and UCP-2 will be recombinant anti- TTC11/FIS1 (ab156865), recombinant anti-DRP1 (ab184247), anti-mitofusin 1 antibody-N-terminal (ab191853), recombinant anti-mitofusin 2 (ab205236), recombinant anti-OPA1 (ab157457), anti-UCP1 (ab155117), and anti-UCP2 (ab247184), respectively.
Mitochondrial reactive oxygen species production | Before and after 12 week supervised exercise program
  Mitochondrial reactive oxygen species production will be assessed with fluorescent imaging of skeletal muscle biopsy samples treated with H2DCFDA (D399, ThermoFisher), which is validated to detect ROS within cells. The validated mitochondrial targeted antioxidant MitoTempo (SML0737, Sigma-Aldrich) will be used to confirm the presence of mitochondrial ROS. EPR will be used to quantify free radicals such as superoxide.

SECONDARY OUTCOMES:
Metabolic equivalents of task | Immediate
  Metabolic equivalents of task (MET) will be used to quantify exercise dose accumulated over the course of the SET or M-SET session. The MET value (measured by metabolic cart) will be multiplied by the number of minutes exercised during each bout. Session MET/min will be summed to quantify total dose (Exercise intensity).
Physical activity enjoyment scale | Immediate
  Physical activity enjoyment scale is an 18-item measure developed to assess the extent to which an individual enjoys a given physical activity. Ratings span from 1(most enjoyment) to 7 (least enjoyment) and the questionnaire has been extensively validated1. The scale will be given at the end of each exercise session.
Rating of perceived exertion | Immediate
  Rating of perceived exertion will be recorded using the Borg Scale, which ranges from 6 (no exertion) to 20 (maximal exertion) at the end of exercise session.
Physical activity average steps/day | Before and after 12 week supervised exercise program
  Physical activity will be measured with an accelerometer (Actigraph GT3X, Actigraph, FL, USA) placed on subjects' hip for seven days after the intervention but prior to the assessment visit. Average steps/day will be calculated. Accelerometers will be given to patients at their last exercise session prior to the assessment data collection.
Muscle strength | Before and after 12 week supervised exercise program
  Muscle strength will be measured with an isokinetic dynamometer (Biodex 4 Medical Systems, Inc. USA). Peak isokinetic strength (torque) of the ankle and hip of the more symptomatic leg will be measured. Subjects will perform one trial of five repetitions at 60 degrees/second to assess strength.
Acceptability | Before and after 12 week supervised exercise program
  In each intervention group, patients will be interviewed after completing the 12 week intervention. Interviews will provide the potential feasibility of exercise by identifying acceptability (satisfaction, intent to continue participation), perceived demand, and practicality (positive/negative effects).
Maximum cadence/day | Before and after 12 week supervised exercise program
  Physical activity will be measured with an accelerometer (Actigraph GT3X, Actigraph, FL, USA) placed on subjects' hip for seven days after the intervention but prior to the assessment visit. Accelerometers will be given to patients at their last exercise session prior to the assessment data collection. Cadence is the number of steps per minute and the maximum cadence in a 24 hour period will be recorded as the maximum cadence/day.
Muscle endurance | Before and after 12 weeks supervised exercise program.
  Muscle endurance will be measured with an isokinetic dynamometer (Biodex 4 Medical Systems, Inc. USA). Peak isokinetic torque of the ankle and hip of the more symptomatic leg will be measured. Subjects will perform one trial of 15 repetitions at 120 degrees/second to assess endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Iraklis I Pipinos, MD, Principal Investigator — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE
Locations (1):
- Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created for sharing purposes. All the outcomes and results will be published in peer-reviewed journals and conference proceedings. The raw data will be shared in a de identified, anonymized dataset upon request with a written agreement from recipient. Therefore, the recipient will be able to complete follow-up and perform new analyses of the raw data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The de-identified, anonymized dataset will only be shared after the completion of the study and publishing the outcomes in peer-reviewed journals and conference proceedings.
Access Criteria: All data obtained from the research study will be securely stored in a VA Data Repository system. Only the PI and authorized VA personnel will have the access to the data. A de-identified, anonymized dataset will be created for sharing purposes. The study data will be shared upon request for potential future uses with a written agreement from the recipient complying with VA guidelines for data sharing.